CLINICAL TRIAL: NCT00515788
Title: Phase I Study of Temozolomide and Intrathecal DepoCyt in Patients With Neoplastic Meningitis
Brief Title: DepoCyt Plus Temozolomide in Patients With Neoplastic Meningitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to slow accrual with no expansion to additional phase.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Enzon Pharmaceuticals, Inc. (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0135
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Neoplastic Meningitis
Keywords: Neoplastic Meningitis; Leptomeningeal Disease; Temozolomide; Temodar; DepoCyt; Liposomal Cytarabine; Liposomal ara-C
MeSH Terms: conditions — Meningeal Carcinomatosis; Meningeal Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DepoCyt + Temozolomide (Experimental): DepoCyt Starting 50 mg Intrathecal Day 1 every 14 days for 12 weeks (6 treatments), then every 28 days for 40 weeks (10 treatments). Temozolomide 100 mg/m^2 by mouth daily for 7 days every 14 days.
  Interventions: Drug: DepoCyt; Drug: Temozolomide

INTERVENTIONS:
Drug: DepoCyt — Starting dose of 50 mg Intrathecal on Day 1 every 14 days for a total of 12 weeks (6 treatments). After the first 12 weeks, 50 mg Intrathecal on Day 1 every 28 days for 40 weeks (10 treatments).
  Other Names: Liposomal Cytarabine; Liposomal ara-C
Drug: Temozolomide — 100 mg/m^2 (capsules) by mouth daily for 7 consecutive days every 14 days.
  Other Names: Temodar

SUMMARY:
Objectives:

- To determine the safety, tolerability and maximum tolerated dose (MTD) of oral temozolomide using a 7 days on and 7 days off regimen combined with intrathecal liposomal cytarabine (DepoCyt) in patients with neoplastic meningitis from solid tumors and systemic lymphoma.

DETAILED DESCRIPTION:
Liposomal cytarabine is a slow-release formulation of cytarabine or Ara-C. It is designed to slowly release cytarabine to increase exposure of cancer cells to the drug in the treatment of leptomeningeal disease. Temozolomide is a chemotherapy drug that is designed to attach to the DNA of rapidly dividing cells (cancer cells). The cells recognize this and self-destruct.

Tests called an Indium-111 or Technetium 99m-DPTA CSF flow study, where radioactive dye is injected into the CSF, will be done to make sure the CSF flows freely throughout the spinal canal. These are done as part of the screening evaluation. If the flow study is okay, you will be eligible to take part in this study. But if there is a block of the CSF pathway, the area may be treated (usually with radiation) and then you can be re-evaluated and may still be enrolled in the study if a repeat flow study shows that the block has been cleared.

If you have a ventriculoperitoneal (VP) or ventriculoatrial (VA) shunt in place, you will have a shunt closure test in which your shunt system will be closed and you will be monitored for 4 hours for the development of clinical signs of increased intracranial pressure. The shunt closure test is performed to allow for a long enough time for the shunt to be closed after liposomal cytarabine is injected. Researchers want to make sure that the drug will stay in the CSF system long enough to perform its function, without being siphoned off through the shunt.

An Ommaya Reservoir (a small round plastic pouch with a tube that goes into the brain and CSF) will be placed under the scalp by a neurosurgeon before starting therapy if you do not already have one in place. The reservoir will be used to deliver the liposomal cytarabine and to collect samples of CSF when they are needed.

Liposomal cytarabine will be given through the Ommaya Reservoir once every 14 days on Day 1 for a total of 12 weeks (6 treatments). This is called Induction Treatment. After the first 12 weeks, liposomal cytarabine will be given on Day 1 every 28 days for 40 weeks (10 treatments). This is called Maintenance Treatment. If you are not already taking daily dexamethasone, you will begin to take dexamethasone by mouth twice a day on the day before the depocyt starts each course and continuing 5 days after the administration of liposomal cytarabine.

Temozolomide will be taken by mouth once a day for 7 days (Days 1 - 7) every 14 days starting from the second treatment of liposomal cytarabine Day 14. You will take it continuously throughout Induction and Maintenance treatment with liposomal cytarabine. Your doctor may prescribe an anti-nausea medication to be taken 1 hour before taking temozolomide. Your doctor will choose the most appropriate anti-nausea medication for you at that time. You should swallow the temozolomide capsules (usually between 1 and 5) whole and quickly one after the other. You should not chew the temozolomide capsules. If vomiting occurs during the course of treatment, no re-dosing will be done before the next scheduled dose. You should take temozolomide at bedtime and fast (not eat or drink anything except water) for at least 1 hour before each dose and for 1 hour after each dose.

Three (3) participants at a time will be enrolled in the Phase I portion of this study. The first group of participants will receive a certain dose of temozolomide. If this dose is tolerated, then an additional 3 will be treated at this dose. If no more than 1 participant has a severe side effect, then that will be the dose for the Phase II portion of this study.

During the Phase II portion, if a participant has shown the ability to tolerate the first dose level, the next dose may be increased, which will be decided by the treating physician at the next treatment timepoint.

During the study, blood samples (about 1 tablespoon each) for routine tests will be repeated every week during Induction and then every 2 weeks during the Maintenance period. The Gd-MRI of the brain and spine will be repeated at Week 6 and 12 and then every 8 weeks. Within 72 hours of each liposomal cytarabine dosing, vital signs and a physical and neurological exam will be done. CSF will be removed from the Ommaya Reservoir every 2 weeks and through lumbar puncture every 6 weeks during Induction and from the Ommaya Reservoir every 4 weeks and through lumbar puncture every 8 weeks during the Maintenance period to look for cancer cells in the fluid.

Treatment will continue unless the disease gets worse or unacceptable side effects occur. Treatment will be given on an outpatient basis. At the end of the study, vital signs, a complete physical and neurological exam, and routine blood tests (about 1 tablespoon) will be performed. CSF samples for cytology, protein, glucose, and cell count will be taken. The Gd-MRI scan will be repeated. You will be asked to complete a questionnaire about how you are feeling.

After completion of the study, you will have a physical and neurological exam and vital signs and CSF samples collected every 28 days for 3 months and then every 3 months for up to 1 year. If there are any signs of your tumor getting worse or returning, you will have a Gd-MRI.

This is an investigational study. Temozolomide is approved by the FDA for the treatment of some brain tumors and is commercially available. Liposomal cytarabine is authorized for research use only in the treatment of brain tumors. The use of these two drugs together is experimental. About 180 patients will take part in this study. About 18 will be enrolled at UT MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be >/=18 years of age
2. All patients with the exception of those with primary brain tumors, must have histologic diagnosis of systemic malignancy. Patients must have the presence of malignant cells in CSF (+CSF) or clinical signs and symptoms of leptomeningeal disease and radiographic abnormalities without malignant cells identified in the CSF (-CSF). Clinical signs/symptoms include cerebral hemispheric, cranial nerve, and/or spinal cord/root dysfunction.
3. Patients must have Karnofsky performance status of >/=60%. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purposes of the performance score.
4. Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy, before entering the study and must be without significant systemic illness. Patients must not have received any systemic therapy for Leptomeningeal disease (LMD) within 3 wks (6 wks if a nitrosourea), intrathecal chemotherapy within 1 wk, or irradiation within 8 wks prior to treatment on this study. Patients previously receiving craniospinal irradiation must have positive cytology or progression of meningeal disease on MRI scan. Patients must not have received whole brain or focal CNS radiotherapy within 1 wk of treatment.
5. Patients must have a platelet count >/= 75,000/mm(3) and ANC >/= 1500/mm(3) within 72 hours prior to intrathecal DepoCyt and temozolomide treatment.
6. Patients must have adequate liver function, total bilirubin < 2.0 mg%; SGPT < 5 times normal; adequate renal function (serum creatinine </= 1.5 mg); and normal metabolic parameters (serum electrolytes, calcium, magnesium, and phosphorus).
7. All patients or their legal guardians must sign a document of informed consent indicating their awareness of the investigational nature and the risks of this study.
8. Ventricular access devices (e.g. an Ommaya reservoir) are mandatory.

Exclusion Criteria:

1. Patients receiving other therapy (either intrathecal or systemic) designed specifically to treat their leptomeningeal disease are not eligible for this study. However, patients receiving concomitant non-cytotoxic therapy (hormonal or cytostatic therapy) to control systemic disease or bulk CNS disease will be eligible, provided the therapy is not a phase I agent, an agent which significantly penetrates the CSF or an agent known to have serious unpredictable CNS side effects.
2. (1. continued) No other cytotoxic chemotherapies are allowed (non-cytotoxic therapies such as herceptin, tarceva, arimidex etc are allowed at the investigator's discretion). Careful documentation of concurrently administered systemic drugs is required.
3. Patients with clinical evidence of obstructive hydrocephalus or compartmentalization of the CSF flow as documented by radioisotope Indium-(111) (Technetium(99) -DTPA when Indium-(111) unavailable) flow study are not eligible for this protocol. CSF obstruction will be determined by routine nuclear medicine CSF flow study parameters. If patients have evidence of block that is subsequently proven to be relieved after focal XRT, these patients can enroll immediately after repeat flow study shows block to be relieved.
4. Patients with a ventriculoperitoneal (VP) or ventriculoatrial (VA) shunt must have an on/off device in their shunt systems to be eligible for the study. Patients must be able to tolerate shunt closure for >/= 4 hours without development of clinical signs of increased intracranial pressure. Patients unable to tolerate shunt closure for >/= 4 hours will not be eligible for the study.
5. Women of childbearing potential (females who are not surgically sterile or who have had a period in the last 12 months) must have a negative serum pregnancy test and must not be lactating.
6. Patients with any uncontrolled infection (life-threatening infection resistant to treatment after 7 days) are not eligible for this study, except those with HIV and AIDS-related lymphomatous meningitis).
7. Use of any other investigational drug within 7 days prior to study entry. This period should be extended if the patient has received any investigational agent that is known to have delayed toxicities after 7 days or a prolonged half-life.
8. Patients not able to undergo magnetic resonance testing. i.e. pacemaker.
9. Patients may not have had prior treatment with Temozolomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) for the combination of Temozolomide and DepoCyt | 28 days
  The MTD is the dose at which 0/3 or 1/6 participants experience Dose Limiting Toxicity (DLT) with the next higher dose having at least 2/3 or 2/6 participants encountering DLT. MTD based on the assessment of DLT during the first 28 days of treatment on the regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Morris D. Groves, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org